CLINICAL TRIAL: NCT00666367
Title: High Dosis of Vitamin D as Treatment for COPD.
Brief Title: Vitamin D as Treatment for Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Prof. Dr. W. Janssens, Katholieke Universiteit Leuven
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-004755-11; S50722
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2010-12-24 (Estimated); Status verified 2009-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Vitamin D (D-cure) will be administered by monthly oral intake. During a prospective follow-up period of one year, the patients will get the normal care with some additional tests for the study.
  Interventions: Drug: D-cure
- 2 (Placebo Comparator): Placebo will be administered by monthly oral intake. During a prospective follow-up period of one year, the patients will get the normal care with some additional tests for the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: D-cure — 4 ml of D-cure (SMB oral intake) in syringe Exacta-Med Oral Dispenser.
  Other Names: license number: D-cure: 465S37F11
  Arms: 1
Drug: Placebo — 4 ml of Arachidis oleum raffinatum Ph. Eur. in syringe Med Oral Dispenser.
  Other Names: Product number: Arachidis oleum raffinatum: *FA072892*
  Arms: 2

SUMMARY:
This project aims to explore the relationship between Vitamin D deficiency and COPD progression via a prospective randomized placebo-controlled study. For this purpose, study was powered to 120 patients hospitalized with an exacerbation of COPD randomly assigned to a monthly oral dose of Vitamin D versus placebo. Taking into account dropouts, 182 patients are randomized during the course of the study

DETAILED DESCRIPTION:
Principal objective: To define the therapeutic effect of Vitamin D in the chronic maintenance treatment of COPD by means of a prospective randomized placebo-controlled double blind study of 182 patients with a follow-up of at least one year. Primary endpoint is the median time to next exacerbation. Secondary endpoints are total number of exacerbations per group, number of exacerbations per patient per year, percentage of patients with one or more exacerbations per year, days of antibiotics and oral steroids, quality of life, FEV1, muscle force and survival.

Other objectives: First, to investigate the role of local and systemic levels of 25-OHD and 1,25-(OH)2D on the intensity and prevalence of bacterial colonisation, inflammatory markers, proteases and markers of oxidative stress in induced sputa and exhaled air. Second, to explore whether correction of Vitamin D deficiency by the oral supplementation of Vitamin D triggers the VDR-mediated cathelicidin pathway and increases local or systemic concentrations of the natural antimicrobial polypeptide cathelicidin with enhanced eradication of bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of COPD exacerbation
* Smoking history of at least ten pack years
* GOLD stage II, III and IV as assessed by a post-bronchodilator spirometry
* Informed consent

Exclusion Criteria:

* Tiffeneau index >70% or FEV1 >80%
* Hypercalcemia
* Sarcoidosis
* Newly discovered symptomatic osteoporosis (proven by DEXA and RX )
* Active cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
median time to next exacerbation. | 1 year

SECONDARY OUTCOMES:
Total number of exacerbations per group, number of exacerbations per patient per year, percentage of patients with one or more exacerbations per year, days of antibiotics and oral steroids, quality of life, FEV1, muscle force and survival. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, Prof., Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - Katholieke Universiteit Leuven, Leuven, Flanders
  - University hospital Leuven, Leuven, Flanders

REFERENCES:
- [Derived] Serre J, Tanjeko AT, Mathyssen C, Heigl T, Sacreas A, Cook DP, Verbeken E, Maes K, Verhaegen J, Pilette C, Vanoirbeek J, Gysemans C, Mathieu C, Vanaudenaerde B, Janssens W, Gayan-Ramirez G. Effects of repeated infections with non-typeable Haemophilus influenzae on lung in vitamin D deficient and smoking mice. Respir Res. 2022 Mar 2;23(1):40. doi: 10.1186/s12931-022-01962-6. PMID 35236342
- [Derived] Lehouck A, Mathieu C, Carremans C, Baeke F, Verhaegen J, Van Eldere J, Decallonne B, Bouillon R, Decramer M, Janssens W. High doses of vitamin D to reduce exacerbations in chronic obstructive pulmonary disease: a randomized trial. Ann Intern Med. 2012 Jan 17;156(2):105-14. doi: 10.7326/0003-4819-156-2-201201170-00004. PMID 22250141